CLINICAL TRIAL: NCT02979405
Title: Effectivenes of Phenylefrine in Prevention of Hypotension During Spinal Anesthesia for Cesarean Delivery: a Randomised Controlled Trial
Brief Title: Effectiveness of Phenylefrine in Prevention of Hypotension During Spinal Anesthesia for Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Industrial de Santander (Other)
Responsible Party: Principal Investigator, Nelly Johanna Puentes Vega, Principal investigator, Universidad Industrial de Santander
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UIS 2016
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hypotension Drug-Induced
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Experimental): Phenylephrine 40 mcg/min, infusion during 5 minutes
  Interventions: Drug: Phenylephrine
- group 2 (Placebo Comparator): Saline solution 21 cc, infusion during 5 minutes
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — prophylactic infusion of phenylephrine 40 mcg/min
  Other Names: prophylactic Phenylephrine

SUMMARY:
Hypotension in patients who are taken to surgery, is a very frequent complication, when the spinal anesthetical technique is used, associating this with significant adverse effects that can lead to morbidity specially in the obstetric patient. The objective of the study is determine if the phenylephrine used of prophylactic form, achieved to prevent the appearance of hypotension in obstetric patients led to Caesarea under spinal anesthesia.

DETAILED DESCRIPTION:
Worldwide, the caesarean section is one of the surgical procedures most frequently performed, representing a challenge to the anesthesiologist, who must administer anesthesia to the mother with minimal effects in the newborn. For this reason, spinal anesthesia emerges as an important option in the management of the obstetrical patient who is going to be taken to Caesarea. The hypotension, is one of the most frequent events adverse associated to this technical anesthetic, represented a risk of complications both, in the mother as in the fetus, by this reason the anesthesiologist must implement different strategies to treat it when this be present. From there arises the necessity of establishing if the phenylephrine, a drug used to treat hypotension, when is administed prophylactically, allows to avoid this effect. We designed a randomized clinical trial in elderly patients over 18 years who are taken to Caesarea, where they formed two groups of patients, one that will administer a prophylactic infusion of phenylephrine compared with placebo, assessing the incidence of hypotension in the two groups and the adverse events most commonly associated with this.

ELIGIBILITY:
Inclusion Criteria:

* pregnant subjects who are to be delivered to cesarean section under subarachnoid anesthesia
* Gestational age >37 weeks

Exclusion Criteria:

Pregnant subjects with:

* Hipertensive disorders in pregnancy
* Acute fetal distress
* Evidence of placental dysfunction
* History of cardiovascular or cerebrovascular diseases
* hypersensitivity to phenylephrine
* Rejection of the patient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Hypotension | caesarean delivery

SECONDARY OUTCOMES:
heart rate | caesarean delivery
Newborn APGAR | Turn off of the newly born: measured to the 1 and 5 minutes from the birth

OTHER OUTCOMES:
Nausea | surgical procedure
Vomiting | surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hector Meléndez, Dr, Study Director — Universidad Industrial de Santander
Locations (1):
- Clinic materno infaltil San Luis, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No